CLINICAL TRIAL: NCT00753311
Title: A Randomized, Double Blind, Controlled Versus Placebo in Parallel Groups, Study to Evaluate the Efficacy of 10 mg Lyophilized Oral Rizatriptan in the Acute Treatment of Migraine in Patients With Unilateral Trigeminal Autonomic Symptoms.
Brief Title: Rizatriptan in Acute Treatment of Migraine in Patients With Unilateral Trigeminal-autonomic Symptoms.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Piero Barbanti, MD, Head, Headache and Pain Unit, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 50/07ssr-msd01-3407
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Migraine
Keywords: migraine; rizatriptan; unilateral trigeminal autonomic symptoms; Migraine with or without aura
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rizatriptan (Active Comparator): Patients with migraine with and without aura will be enrolled and randomly provided with study drug (rizatriptan 10 mg MLT or placebo, ratio 1:1). Patients were encouraged to take migraine medication as soon as their migraine headache became moderate or severe. If the moderate or severe migraine headache persisted 2 h after dosing, or recurred within 24 h, patients had the option of taking their own rescue medication but triptans and ergot derivatives were prohibited for 24 h after study medication intake.
  Interventions: Drug: rizatriptan or placebo
- placebo (Placebo Comparator): Patients who met all the study entry criteria were enrolled and randomly allocated to receive either rizatriptan 10 mg wafer or placebo (ratio 1:1).Patients were encouraged to take migraine medication as soon as their migraine headache became moderate or severe. If the moderate or severe migraine headache persisted 2 h after dosing, or recurred within 24 h, patients had the option of taking their own rescue medication but triptans and ergot derivatives were prohibited for 24 h after study medication intake.
  Interventions: Drug: rizatriptan or placebo

INTERVENTIONS:
Drug: rizatriptan or placebo — Patient took 1 rizatriptan 10 mg wafer or placebo as soon as their migraine headache became of moderate or severe intensity.

SUMMARY:
Triptans are first choice drugs in the acute treatment of migraine and cluster headache. However, while in cluster headache the response rate to subcutaneous sumatriptan is 96%, around 30% of patients fail to respond to a particular triptan. Nonresponse is likely to be due to a variety of factors, including low and inconsistent absorption, inadequate dosing, and variability in individual response5. Timing of administration is also a crucial issue. In fact, an early treatment of the attack, when the pain is still mild, may increase the responders rate by circumventing the development of cutaneous allodynia (expression of central sensitization of pain pathway) during the course of the attack.

Several studies have been performed in an attempt to genetically, psychologically and clinically characterize the triptan responders but failed to provide conclusive results.

Nevertheless, we suggested that the presence of UAs during the migraine attack might predict a good response to triptans. UAs are common in migraine patients. They have been reported in almost one out of two migraineurs (45.8%) attending a tertiary headache centre and in more than one out of four (26.9%) in a population-based study. In an open study with sumatriptan 50 mg performed on 72 migraine patients with UAs, we described pain relief in 65.3% of the patients at 1 h and in 81.9% at 2 h, while pain-free in 30.6% at 1 h and in 61.1% at 2 h. We hypothesized a large-scale recruitment of peripheral neurovascular 5-HT1B/1D receptors consequent to the activation of the trigeminal-autonomic reflex in such patients. Our hypothesis has received further confirmation by the demonstration of higher levels of calcitonin gene-related peptide, neurokinin A and vasoactive intestinal peptide (the hallmark of the activation of the trigeminal autonomic reflex) in external jugular blood in rizatriptan responders than in non-responders.

The investigators therefore postulate that migraineurs with UAs may respond better to rizatriptan than "general" migraine population.

The aim of the study is to evaluate the efficacy of rizatriptan 10 mg lyophilized wafer (MLT) compared to placebo in the treatment of acute migraine in patients with unilateral autonomic symptoms (UAs: unilateral lacrimation, eye redness, eyelid oedema, nasal congestion or rhinorrhoea, miosis or ptosis, forehead or facial sweating) during the migraine attack.

DETAILED DESCRIPTION:
We tested the hypothesis that the presence of unilateral cranial autonomic symptoms in migraine predicts a good response to triptans. In this randomized, double-blind, placebo-controlled study 80 migraineurs with unilateral cranial autonomic symptoms were assigned to rizatriptan 10 mg wafer or placebo (ratio 1:1) and treated for a single moderate or severe migraine attack. The primary endpoints were pain freedom at 2 h and total migraine freedom at 2 h. Secondary endpoints included pain relief, no associated symptoms and sustained pain freedom or relief. Significantly more patients reported pain freedom at 2 h after taking rizatriptan than after placebo (54% vs 8%; p<0.001). Similarly, significantly more patients reported total migraine freedom at 2 h after rizatriptan than after placebo (51% vs 8%; p<0.001). Rizatriptan was also more effective than placebo on most secondary endpoints. Migraineurs with unilateral cranial autonomic symptoms respond better than the general migraine population to rizatriptan, probably owing to intense trigeminal peripheral afferent activation which strongly recruits peripheral neurovascular 5-HT1B/1D receptors. Acute and preventive pharmacological trials in migraine should focus also on this subset of migraine patients.

ELIGIBILITY:
Inclusion Criteria:

Male or female ≥18 years of age at screening. History of migraine with or without aura > 1 year with ≥1 and ≤8 moderate or Severe migraine attacks per month in the 2 months prior to screening that typically last longer than 2 hours.During the migraine attack (if untreated) patient has every time at least 1 of the following symptoms due to the activation of the trigeminal-autonomic reflex (UAs): unilateral conjunctival injection and/or lacrimation and/or nasal congestion/rhinorrhea and/or ptosis and/or eyelid oedema and/or forehead/facial sweating. A patient who is of reproductive potential agrees to remain abstinent or use (or have their partner use) 2 acceptable methods of birth control within the projected duration of the study (intrauterine device (IUD),diaphragm with spermicide,contraceptive sponge,condoms,vasectomy.Health condition in the opinion of the investigator based on screening assessment including medical history,physical examination,and laboratory testing carried out within ~2 months prior to study treatment.Patient agrees to participate by giving written informed consent and able to complete the study questionnaire(s)and paper diary.

Exclusion Criteria:

Patient is pregnant or breast-feeding, or expecting to conceive within the projected duration of the study.Patient has difficulty distinguishing his/her migraine attacks from tension or interval headaches.History of predominantly mild migraine attacks or migraines usually resolved spontaneously in less than 2 hours.Basilar or hemiplegic migraine headache.Patient has more than 15 headache-days per month or has taken medication for acute headache on more than 10 days per month in any of the 3 months prior to screening.Patient is taking migraine Propranolol or has discontinued it from less than 14 days.Patient is taking migraine prophylactic medication where the prescribed daily dose has changed during the 3 months prior to screening.Patient was > 50 years old at age of migraine onset. Recent history (within the past 5 years) or current evidence of drug or alcohol abuse or is a "recreational user" of illicit drugs.Concomitant use of propranolol, ergot derivatives, methysergide or MAO inhibitors.Hypersensitivity to any marketed 5HT1B/1D receptor agonist.History or clinical evidence of ischemic heart disease (e.g., angina pectoris of any type, history of myocardial infarction or documented silent ischemia) or symptoms or findings consistent with ischemic heart disease, coronary artery vasospasm (including Prinzmetal's variant angina,or other significant underlying cardiovascular disease.Patient has clinical,laboratory,or ECG evidence of uncontrolled hypertension, uncontrolled diabetes, or significant pulmonary, renal, hepatic, endocrine, or other systemic disease in the opinion of the investigator.Patient has, in the opinion of the investigator, other confounding pain syndromes, psychiatric conditions such as uncontrolled major depression based on criteria such as DSM-IV, dementia or significant neurological disorders other than migraine.History of neoplastic disease ≤ 5 years prior to signing informed consent.Patient has a history of gastric or small intestinal surgery (including gastric bypass surgery or banding), or has a disease that causes malabsorption. History or current evidence of any clinically significant disease that according to the investigator might confound the results of the study, complicate the interpretation of the study results, interfere with the patient's participation for the full duration of the study, or pose an additional undue risk to the patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Rating of headache severity at baseline and 2 hours postdose. | 12 months

SECONDARY OUTCOMES:
Rating of headache severity, associated symptoms and disability at 0.5, 1, 1.5, 2, 3, 4, and 24 hours post dose. b.Headache recurrence. c.Use of rescue medication. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Piero Barbanti, MD, PhD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele Pisana, Clinical Trial Center, Rome, Italy

REFERENCES:
- [Derived] Barbanti P, Fofi L, Dall'Armi V, Aurilia C, Egeo G, Vanacore N, Bonassi S. Rizatriptan in migraineurs with unilateral cranial autonomic symptoms: a double-blind trial. J Headache Pain. 2012 Jul;13(5):407-14. doi: 10.1007/s10194-012-0440-y. Epub 2012 Mar 30. PMID 22460943